CLINICAL TRIAL: NCT07318454
Title: A Randomized Controlled Trial Comparing Abdominal Expansion and Abdominal Drawing-In Training With Manual and Verbal Cueing in Individuals With Chronic Non-Specific Low Back Pain
Brief Title: Comparison of Abdominal Expansion and Abdominal Drawing-In Training With Manual and Verbal Cueing in Chronic Non-Specific Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Wendy Tzyy-Jiuan Wang, Professor, Department of Physical Therapy, National Yang Ming Chiao Tung University, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NYCU114229AE-S3
Record Dates: First submitted 2025-12-23; First posted 2026-01-06 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Chronic Low Back Pain (Non-specific, Uncomplicated)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ADIM With Verbal Cueing (Experimental): Participants receive abdominal drawing-in manoeuvre training with verbal cueing, delivered twice weekly for 4 weeks.
  Interventions: Behavioral: Abdominal Drawing-In Manoeuvre Training
- ADIM With Manual Cueing (Experimental): Participants receive abdominal drawing-in manoeuvre training with manual facilitation, delivered twice weekly for 4 weeks.
  Interventions: Behavioral: Abdominal Drawing-In Manoeuvre Training
- DNS-AE With Verbal Cueing (Experimental): Participants receive Dynamic Neuromusculoskeletal Stabilization abdominal expansion training with verbal cueing, delivered twice weekly for 4 weeks.
  Interventions: Behavioral: Dynamic Neuromusculoskeletal Stabilization Abdominal Expansion Training
- DNS-AE With Manual Cueing (Experimental): Participants receive Dynamic Neuromusculoskeletal Stabilization abdominal expansion training with manual facilitation, delivered twice weekly for 4 weeks.
  Interventions: Behavioral: Dynamic Neuromusculoskeletal Stabilization Abdominal Expansion Training

INTERVENTIONS:
Behavioral: Abdominal Drawing-In Manoeuvre Training — Abdominal drawing-in manoeuvre (ADIM) training is a core stability exercise strategy emphasizing selective activation and coordination of the deep abdominal musculature to enhance local trunk stability. Participants receive individualized, one-on-one training delivered by licensed physical therapists, conducted twice weekly for 4 weeks. Training is performed across functional positions and task-specific movements, with instruction provided using either verbal cueing or manual facilitation according to group allocation.
  Arms: ADIM With Manual Cueing; ADIM With Verbal Cueing
Behavioral: Dynamic Neuromusculoskeletal Stabilization Abdominal Expansion Training — Dynamic Neuromusculoskeletal Stabilization abdominal expansion (DNS-AE) training focuses on coordinated breathing and abdominal expansion to facilitate intra-abdominal pressure regulation and integrated postural control. Participants receive individualized, one-on-one training delivered by licensed physical therapists, conducted twice weekly for 4 weeks. Training is performed across functional positions and task-specific movements, with instruction provided using either verbal cueing or manual facilitation according to group allocation.
  Arms: DNS-AE With Manual Cueing; DNS-AE With Verbal Cueing

SUMMARY:
This study aims to investigate the interactive effects of two core stability training strategies-abdominal drawing-in manoeuvre (ADIM) and Dynamic Neuromusculoskeletal Stabilization abdominal expansion (DNS-AE)-and two instructional approaches (verbal cueing and manual facilitation) on training outcomes in individuals with chronic non-specific low back pain.

A 2×2 factorial randomized controlled trial design will be employed. Ninety-six participants with chronic non-specific low back pain will be randomly allocated, using block randomization, to one of four intervention groups in equal proportions. All groups will receive a 4-week intervention program, with training conducted twice per week.

Outcome measures will be assessed at four time points: before the intervention (baseline), immediately after the first training session, at the completion of the 4-week intervention, and at a 3-month follow-up, to evaluate short-term and mid-term effects as well as the sustainability of training outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Clinically diagnosed with chronic non-specific low back pain, with symptoms persisting for more than 12 weeks.
* Able to understand the study procedures and comply with the full intervention and assessment protocol.

Exclusion Criteria:

* History of surgery involving the lower back or lower extremities.
* Presence of neurological symptoms, such as numbness or tingling sensations.
* Signs or symptoms of nerve root compression.
* History of any surgical procedure within the past 3 months.
* Diagnosis of cancer.
* Presence of major medical or psychiatric disorders.
* Presence of systemic inflammatory disease.
* Pregnancy.
* Structural scoliosis of the spine.
* Inability to ambulate or stand independently, or other conditions deemed unsuitable for participation.
* Participation in any movement control-based exercise training within the past year.
* Accumulated experience of more than 4 weeks of abdominal drawing-in manoeuvre (ADIM) training or Dynamic Neuromusculoskeletal Stabilization abdominal expansion (DNS-AE) training within the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | At baseline, after the first week of intervention, and at the end of the 4-week intervention.
  Pain intensity assessed using the Visual Analogue Scale (VAS), ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable, with higher scores indicating greater pain intensity.
Movement control performance | At baseline, after the first week of intervention, and at the end of the 4-week intervention.
  Movement control performance assessed using the Nine-Item Movement Control Test Battery, which evaluates movement quality during standardized functional movement tasks. Each item is scored according to predefined error-based criteria, and item scores are summed to produce a total score ranging from 0 to 93, with higher scores indicating poorer movement control performance.

SECONDARY OUTCOMES:
Disability related to low back pain | At baseline, at the end of the 4-week intervention, and at 3-month follow-up.
  Disability assessed using the Oswestry Disability Index (ODI), with total scores ranging from 0 %to 100%, where higher scores indicate greater disability.
Patient-specific functional ability | At baseline, at the end of the 4-week intervention, and at 3-month follow-up.
  Functional ability assessed using the Patient-Specific Functional Scale (PSFS), with scores ranging from 0 to 10, where 0 indicates inability to perform the activity and 10 indicates the ability to perform the activity at the pre-injury or normal level, with higher scores indicating better functional ability.
Perceived movement difficulty assessed using the Perceived Difficulty Index (PDI). | At baseline, after the first week of intervention, and at the end of the 4-week intervention.
  Perceived difficulty during movement performance assessed using the Perceived Difficulty Index (PDI). Participants rate the level of difficulty experienced during the movement tasks on a numeric rating scale ranging from 0 to 10, where 0 indicates no perceived difficulty and 10 indicates extreme difficulty, with higher scores indicating greater perceived difficulty.
Central sensitization symptoms | At baseline and at the end of the 4-week intervention.
  Symptoms related to central sensitization assessed using the Central Sensitization Inventory (CSI), with total scores ranging from 0 to 100, where higher scores indicate greater symptom severity related to central sensitization.
Fear-avoidance beliefs | At baseline and at the end of the 4-week intervention.
  Fear-avoidance beliefs assessed using the Fear-Avoidance Beliefs Questionnaire (FABQ), with total scores ranging from 0 to 96, where higher scores indicate greater fear-avoidance beliefs.
Pain catastrophizing | At baseline and at the end of the 4-week intervention.
  Pain catastrophizing assessed using the Pain Catastrophizing Scale (PCS), with total scores ranging from 0 to 52, where higher scores indicate greater pain catastrophizing.
Pressure pain threshold | At baseline and at the end of the 4-week intervention.
  Pressure pain threshold (PPT) assessed using a pressure algometer.
Global perceived change | At the end of the 4-week intervention and at 3-month follow-up.
  Overall perceived change assessed using the Global Rating of Change (GROC) scale, ranging from -7 to +7, where negative scores indicate perceived worsening, 0 indicates no change, and positive scores indicate perceived improvement, with higher scores indicating greater perceived improvement.
Learning acquisition during training | After each training session during the 4-week intervention.
  Learning acquisition assessed by the instructor after each training session using a numeric rating scale from 0 to 10.